CLINICAL TRIAL: NCT00012844
Title: Redesigning Patient Handling Tasks to Prevent Nursing Back Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NRI 95-150
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Back Pain; Occupational Diseases
Keywords: Musculoskeletal Disorders; Patient Lifting; Occupational Accidents
MeSH Terms: conditions — Back Pain; Occupational Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Device: Redesigning patient handling tasks using equip: Arjo Bianca Overhead Lift, Hill-Rom Resident Transfer Device, TranSit Chair, Total Care Bed; Procedure: Redesigned patient handling tasks using work practice controls: setting bed height at correct level; applying anti-embolism stockings from foot of bed

INTERVENTIONS:
Device: Redesigning patient handling tasks using equip: Arjo Bianca Overhead Lift, Hill-Rom Resident Transfer Device, TranSit Chair, Total Care Bed
Procedure: Redesigned patient handling tasks using work practice controls: setting bed height at correct level; applying anti-embolism stockings from foot of bed

SUMMARY:
This study is one of several initiated by the investigators to reduce musculoskeletal injuries in patient care providers. Nurses have one of the highest incidences of work related back injuries of any profession. Over the past 20 years, efforts to reduce work-related injuries in nursing have been largely unsuccessful.

DETAILED DESCRIPTION:
Background:

This study is one of several initiated by the investigators to reduce musculoskeletal injuries in patient care providers. Nurses have one of the highest incidences of work related back injuries of any profession. Over the past 20 years, efforts to reduce work-related injuries in nursing have been largely unsuccessful.

Objectives:

The goal of this study is to reduce the incidence and severity of occupational musculoskeletal injuries in nursing through the redesign of stressful patient handling tasks. This study addresses three objectives: 1) conduct a quantitative, biomechanically based, ergonomic evaluation of the eleven "at risk" tasks in nursing practice; 2) redesign the techniques or equipment needed to perform these tasks safely or with reduced risk of musculoskeletal injury; and 3) conduct laboratory- based assessment of the biomechanical benefit of the proposed intervention strategies.

Methods:

Using a randomized experimental design with a control group, ten "at risk" tasks will be evaluated. The sample included 160 experienced nursing staff. Data were collected using: 1) Caregiver Data Form and Anthropometry Data Sheet; 2) 3-D Electromagnetic Tracking System; 3) EMG; and 4) modified Borg Scale for Perceived Comfort. Include: caregiver characteristics, joint torque, spinal forces, spinal tolerance limit and damage load limit, erector spinae surface EMG, joint angles, percent of population capable of performing each task by gender, velocity of lift, reach, heart rate, and perceived comfort.

Status:

This project is complete.

ELIGIBILITY:
Inclusion Criteria:

Subjects included RNs, LPNs, and Nas with a minimum of 6 months experience and a job description that included a minimum of 80% direct patient care responsibilities. Subjects were required to be injury free for at least one year, as evidenced by a brief orthopedic examination and interview. The orthopedic evaluation included an examination of posture, gait, range of motion, sensory deficits, muscle exam, and straight leg raise. We excluded subjects with self-report of injury or any positive finding of back musculoskeletal disorders within the past 12 months.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Study Completion 1999-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L. Nelson, RN PhD FAAN, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States